CLINICAL TRIAL: NCT02962973
Title: Clinical Evaluation of the Carmat Total Artificial Heart for Patients With Advanced Heart Failure
Brief Title: European Clinical Evaluation of the Carmat Total Artificial Heart
Acronym: ADVANCEHF
Status: Suspended | Phase: Not Applicable | Type: Interventional
Sponsor: Carmat SAS (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CAR2016-01; CIV-FR-16-09-016865 (Other: EUDAMED)
Record Dates: First submitted 2016-11-08; First posted 2016-11-15 (Estimated); Last update posted 2025-02-14 (Actual); Status verified 2025-02

CONDITIONS: Advanced Heart Failure
Keywords: Advanced heart failure; Total artificial heart
MeSH Terms: interventions — Surgical Procedures, Operative

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Carmat TAH (Experimental): The surgical intervention takes place through a midsternotomy utilizing cardiopulmonary bypass. The device is then connected via a percutaneous driveline to an external controller and batteries and takes over the circulation.
  Interventions: Device: CARMAT TAH; Procedure: Surgical intervention

INTERVENTIONS:
Device: CARMAT TAH
Procedure: Surgical intervention

SUMMARY:
The objective of this clinical investigation is to evaluate the safety and performance of the Carmat Total Artificial Heart (TAH) in subjects with advanced heart failure requiring biventricular support.

Each subject receiving the Carmat TAH will be evaluated at 6 months (180 days) for primary and secondary endpoints with further follow-up assessments up to 2 years.

The results of the study will be used to support a CE mark application.

DETAILED DESCRIPTION:
Center selection is based on the following: experience with VAD/TAH implantation and record of good results in this patient population (% of survival), the infrastructure required to perform the clinical investigation (especially the surgical and cardiology teams); site resources and experience to manage the clinical study and the patient population; the adherence to the standards of Good Clinical Practice. A specific focus during the site selection is done on dedicated VAD - nurse team to ensure that:

* Sites are experienced in the selection of patients whom require a mechanical circulatory support. Social and psychological conditions of the patient and family must be considered to ensure patient and family commitment in the care pathway,
* Close supervision of patients on the use of the device (when changing batteries) by experienced hospital professionals is guarantee;
* Extensive hospital training program and regular support for patients and family - relatives are ensured.

ELIGIBILITY:
Inclusion Criteria:

1. Patient age: 18 to 75 years
2. Inotrope dependent or cardiac Index (CI) < 2.2 L/min/m2 if inotropes are contra-indicated (heart failure due to restrictive or constrictive physiology).
3. On Optimal Medical Management as judged by the investigator based on current Heart Failure practice guidelines (ESC/AHA)
4. Eligible to biventricular Mechanical Circulatory Support according to ISHLT guidelines for mechanical circulatory support:

   1. Biventricular failure with at least two of the following hemodynamic/ echocardiographic measurements implying right heart failure:

      1. RVEF ≤ 30%
      2. RVSWI ≤ 0.25 mmHg*L/m2
      3. TAPSE ≤ 14mm
      4. RV-to-LV end-diastolic diameter ratio > 0.72
      5. CVP > 15 mmHg
      6. CVP-to-PCWP ratio > 0.63
      7. Tricuspid insufficiency grade 4
   2. Treatment-refractory recurrent and sustained ventricular tachycardia or ventricular fibrillation in the presence of untreatable arrhythmogenic pathologic substrate
   3. Heart failure due to restrictive or constrictive physiology (e.g., hypertrophic cardiomyopathy, cardiac amyloidosis / senile or other infiltrative heart disease)
5. Anatomic compatibility confirmed using 3D imaging (CT-scan)
6. Patient's affiliation to health care insurance, if local requirement
7. Patient has signed the informed consent and committed to follow study requirements

Exclusion Criteria:

1. Body Mass Index (BMI) < 15 or > 47
2. Existence of any ongoing non-temporary mechanical circulatory support
3. Existence of any temporary mechanical circulatory support other than IABP and Impella
4. History of cardiac or other organ transplant
5. Patients who have required cardiopulmonary resuscitation for > 30 minutes within 14 days prior to implant
6. Known intolerance to anticoagulant or antiplatelet therapies
7. Coagulopathy defined by platelets < 100k/μl or INR ≥ 1.5 not due to anticoagulant therapy
8. Cerebro-vascular accident < 3 months or symptomatic or a known > 80% carotid stenosis
9. Known abdominal or thoracic aortic aneurysm > 5 cm
10. End-organ dysfunction as per investigator judgment and following but not limited criteria:

    1. Total bilirubin > 100 μmol/L (5,8 mg/dl) or cirrhosis evidenced by ultrasound, CT-scan or positive biopsy
    2. GFR < 30ml/min/1.73m2
11. History of severe Chronic Obstructive Pulmonary Disease or severe restrictive lung disease
12. Recent blood stream infection (<7 days)
13. Documented amyloid light-chain (AL amyloidosis)
14. Hemodynamically significant peripheral vascular disease accompanied by rest pain or extremity ulceration
15. Illness, other than heart disease, that would limit survival to less than 1 year
16. Irreversible cognitive dysfunction, psychosocial issues or psychiatric disease, likely to impair compliance with the study protocol and TAH management
17. Participation in any other clinical investigation that is likely to confound study results or affect the study
18. Pregnancy or breast feeding (woman in age of childbearing will have to show negative pregnancy test)

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2016-09 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
Proportion of participants with survival at 180 days | 180 days
  Success is defined as survival at 180 days after Carmat TAH implantation or transplanted if before 180 days.

SECONDARY OUTCOMES:
Overall survival | 180 days
  Patient follow-up
General health status change (1) | 180 days
  Measured with the EuroQol EQ-5D questionnaire, a descriptive system of health-related quality of life states consisting of five dimensions (mobility, self-care, usual activities, pain/discomfort, anxiety/depression) each of which can take one of five responses (EQ-5D-5L). The responses record five levels of severity (1:no problems; 2:slight problems; 3:moderate problems 4:severe problems; 5:extreme problems) within a particular EQ-5D dimension.
General health status change (2) | 180 days
  Change as measured by the SF-36 questionnaire, consisting of eight scaled scores, which are the weighted sums of the questions in their section. Each scale is directly transformed into a 0-100 scale on the assumption that each question carries equal weight. The lower the score the more disability.
Functional status change | 180 days
  New York Heart Association (NYHA) functional classification (regression scale I, II, III, IV)
Change in functional status measured by the Six Minutes Walk Test | 180 days
  The 6-min walk test is a submaximal exercise test that entails measurement of distance walked over a span of 6 minutes. The 6-minute walk distance provides a measure for integrated global response of multiple cardiopulmonary and musculoskeletal systems involved in exercise.
Adverse events | 180 days
  Adverse Event Rates will be captured per the INTERMACS definitions
hospital readmission rate | 180 days
  Rate of unplanned readmissions to the hospital
  * Frequency and incidence of all adverse events
  * Frequency and incidence of pre-defined anticipated adverse events
  * Frequency, incidence and type of device malfunction

CONTACTS AND LOCATIONS:
Overall Officials: Piet Jansen, MD, PhD, Study Director — Carmat SAS
Locations (2):
- "National Research Cardiac Surgery Center", Astana, Kazakhstan
- UMC Utrecht, Utrecht, Netherlands

REFERENCES:
- [Derived] Netuka I, Pya Y, Bekbossynova M, Ivak P, Konarik M, Gustafsson F, Smadja DM, Jansen P, Latremouille C. Initial bridge to transplant experience with a bioprosthetic autoregulated artificial heart. J Heart Lung Transplant. 2020 Dec;39(12):1491-1493. doi: 10.1016/j.healun.2020.07.004. Epub 2020 Jul 14. No abstract available. PMID 32758387
- [Derived] Bizouarn P, Roussel JC, Trochu JN, Perles JC, Latremouille C. Effects of pre-load variations on hemodynamic parameters with a pulsatile autoregulated artificial heart during the early post-operative period. J Heart Lung Transplant. 2018 Jan;37(1):161-163. doi: 10.1016/j.healun.2017.06.018. Epub 2017 Jul 8. No abstract available. PMID 28736110